CLINICAL TRIAL: NCT05463783
Title: Effect of Darunavir/Cobicistat/Emtricitabine/Tenofovir Alafenamide and Bictegravir/Emtricitabine/Tenofovir Alafenamide on the Circulatory microRNA Profile in Treatment naïve HIV Patients, and Its Correlation With Change in Body Weight
Brief Title: Effect of Biktarvy & Symtuza on microRNAs in HIV and Correlation With Weight Gain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: East Carolina University (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Principal Investigator, Paul Cook, Clinical Professor, East Carolina University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UMCIRB 22-000833
Record Dates: First submitted 2022-05-25; First posted 2022-07-19 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections; Obesity
Keywords: microRNA; miRNA; ARV; Antiretroviral medications
MeSH Terms: conditions — HIV Infections; Obesity | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination; symtuza; Darunavir

STUDY DESIGN:
Intervention Model Description: Interventional, open-label, parallel-group, randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biktarvy (Experimental): 15 subjects will get Biktarvy (single-tablet regimen of bictegravir/emtricitabine/tenofovir alafenamide) once daily.
  Interventions: Drug: Biktarvy
- Symtuza (Experimental): 15 subjects will get Symtuza (single-tablet regimen of darunavir/cobicistat/emtricitabine/tenofovir alafenamide) once daily.
  Interventions: Drug: Symtuza

INTERVENTIONS:
Drug: Biktarvy — microRNA profiles of subjects on Biktarvy, will be compared with those who are on Symtuza, at various time points.
  Other Names: bictegravir/emtricitabine/tenofovir alafenamide
  Arms: Biktarvy
Drug: Symtuza — microRNA profiles of subjects on Symtuza, will be compared with those who are on Biktarvy, at various time points.
  Other Names: darunavir/cobicistat/emtricitabine/tenofovir alafenamide
  Arms: Symtuza

SUMMARY:
The purpose of this research study is to understand why certain HIV medication regimens (called anti-retroviral or ARV medications) cause more weight gain than others. In this research, the investigators will compare micro-RNA profiles of people who take Symtuza(darunavir(D)/cobicistat(C)/emtricitabine(F)/tenofovir alafenamide (TAF))[D/C/F/TAF] with those who take Biktarvy(bictegravir(B)/emtricitabine(F)/tenofovir alafenamide (TAF))[B/F/TAF] and try to correlate this with the change in body weight and BMI over a course of 48 weeks. The investigators will also attempt to monitor the calorie intake of the participants in the two groups and correlate it with treatment-induced weight gain. Micro-RNAs are small molecules that are produced naturally in the human body, and which are responsible for modifying the expressions of genes. They have the potential to be used in diagnostic and therapeutic medicine and their putative role has been explored in many diseases across many clinical trials. By doing this research, the investigators hope to learn more about their role in HIV disease and its correlation with treatment-induced weight gain.

DETAILED DESCRIPTION:
With advances in HIV treatment, the life expectancy of persons with HIV (PWH) has improved and complications associated with antiretroviral (ARV) medications have become more apparent. Among them, weight gain and obesity, because of their associated complications, is one of the more concerning ones. Certain drug regimens are more adipogenic than others, but not a lot is known about molecular mechanisms responsible for these differences. Micro RNAs (miRNAs) are small non-coding RNAs that control gene expression and regulate a wide array of biological processes. In recent years miRNAs have been studied in a number of diseases for diagnostic and even therapeutic purposes. There are studies showing differences in miRNA profiles in obese vs non-obese non-HIV population, as well as certain miRNAs as biomarkers of response to weight-loss diets. In PWH, there are studies that looked at the effect of HIV infection on the miRNA profile and how a particular miRNA profile is predictive of ARV resistance. But there are no studies that specifically looked at how ARV medications alter the miRNA profile and how (in terms of miRNA profiles) one combination is more adipogenic than the other.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects age >/=18 years
2. HIV infection with HIV RNA >/= 1000 copies/ml of plasma
3. Treatment naïve
4. Have access to a smartphone with internet access
5. Willing to provide written informed consent.

Exclusion Criteria:

1. Morbid obesity (BMI>/=40) or cachexia (BMI=/<20)
2. Known or suspected active substance abuse that in the opinion of the investigator would impact study participation
3. On medications associated with weight loss or gain, including insulin, glucagon-like peptide(GLP)-1 analogs, anti-depressants, antipsychotics, corticosteroids, orlistat
4. Bedbound due to other chronic conditions
5. Pregnant females
6. Prisoners
7. Unwilling or unable to comply with protocol requirements.
8. On medication known to interact significantly with any of the components of Symtuza or Biktarvy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
miRNA(microRNA) profiles of the two groups | 48 weeks
  we will monitor microRNAs of the two groups
Change from baseline in Body mass index-BMI(kg/m^2) of the participants | 48 weeks
  Weight(in kilograms or kg) and height(in meters or m) will be combined to report BMI in kg/m^2
Change from baseline in body weight(in kilograms or kg) of the participants | 48 weeks
  we will monitor change in body weight & BMI

SECONDARY OUTCOMES:
Calorie intake of subjects in the two groups. | 48 weeks
  we will monitor calorie intake of subjects in two grouos

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cook, MD, Principal Investigator — East Carolina University
Locations (1):
- Adult Specialty Care Clinic-East Carolina University, Greenville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No